CLINICAL TRIAL: NCT02215928
Title: Tumor Genomic Profiling: A Personalized Medicine Approach
Brief Title: Genomic Profiling in Recommending Treatment for Patients With Metastatic Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-29525; NCI-2014-01662 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — liquid biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (tumor genomic profiling): Tissue samples are collected at baseline and blood for liquid biopsy is collected at baseline and every 6-8 weeks during active treatment. Tissue samples are analyzed via sequencing for tumor genomic profiling.
  Interventions: Genetic: mutation analysis; Other: cytology specimen collection procedure; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: mutation analysis — Correlative studies
Other: cytology specimen collection procedure — Correlative studies
  Other Names: cytologic sampling
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies using genomic profiling to recommend anticancer treatment to patients with cancer that has spread beyond the original site of the tumor (metastatic cancer). Genomic profiling studies the deoxyribonucleic acid (DNA) of a tumor to detect genetic changes or abnormalities. This information can then be used to recommend treatments that may be more likely to result in a beneficial response. It is not yet known whether genomic profiling will detect abnormalities that can be used to make treatment recommendations and whether treatment based on genomic profiling is more effective than standard treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility of integrating tumor genomic profiling in the adult oncology clinic at the Stanford Cancer Institute.

SECONDARY OBJECTIVES:

I. Determine the percentage of tumors that harbor "actionable" genomic changes. II. Explore effects of individual molecular profiling including the percent of time that profiling changes the treatment.

III. Determine the number of cases in which a genomically identified targeted therapy is available.

IV. Determine the clinical benefit of genomic based therapy, as defined by: response rate (according to Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 response criteria); the percent of patients with non-progression at 4 months, and overall survival, in patients whose therapy is selected based on profiling.

V. Determine if circulating free tumor DNA (ctDNA) in the blood stream (liquid biopsy) yields similar genomic results as the metastatic tumor analysis.

VI. Determine if ctDNA analysis during treatment correlates with RECIST 1.1 criteria in predicting response.

OUTLINE:

Tissue samples are collected at baseline and blood for liquid biopsy is collected at baseline and every 6-8 weeks during active treatment. Tissue samples are analyzed via sequencing for tumor genomic profiling.

After completion of active treatment, participants are followed up at 4, 8, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Understand and provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization prior to initiation of any study-specific procedures
* Have a diagnosis of metastatic, incurable cancer and have progressed on at least one line of systemic therapy OR a cancer with no standard 1st-line systemic therapy shown to prolong survival (or where a clinical trial recommended as the 1st-line option)
* Measurable disease (RECIST 1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* In the opinion of the investigator, be medically suitable for and willing to undergo a biopsy or surgical procedure to obtain tissue as a part of routine care for their malignancy OR have adequate archival tissue from a previous biopsy available for profiling
* Female patients of childbearing potential must have a negative pregnancy test and agree to use at least one form of contraception during the study and for at least one month after treatment discontinuation; for the purposes of this study, child-bearing potential is defined as: all female patients that were not in post-menopause for at least one year or are surgically sterile
* Male patients must use a form of barrier contraception approved by the investigator/treating physician during the study and for at least one month after treatment discontinuation

Exclusion Criteria:

* Have lesions that are not accessible to biopsy or not planned for biopsy as part of routine care OR if archival tissue will be used for profiling, an insufficient amount is available
* Have diagnosis of a hematologic malignancy
* Have symptomatic central nervous system (CNS) metastasis; patients with a history of CNS metastases who have been treated with whole brain irradiation must be stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on a stable dose of steroids for >= 2 weeks prior to enrollment
* Have uncontrolled concurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent
* Have known human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) infection
* Are pregnant or breast-feeding patients or any patient with childbearing potential not using adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult oncology clinic at the Stanford Cancer Institute
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-07-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility, measured as the proportion of patients with at least one actionable alteration | Baseline
  An actionable alteration is defined as availability of targeted therapy, scored as: A) an FDA-approved drug, B) an FDA-approved drug in another tumor type, or C) a drug that is not yet approved but has a clinical trial open. The percentage of patients in the "profile" arm with successful profiling will be calculated and further characterized by availability category.

SECONDARY OUTCOMES:
Drugs (if any) that target alterations found in a patient's tumor material at baseline, as identified by the Molecular Tumor Board | Baseline
Drugs (if any) that target alterations found in a patient's peripheral blood at baseline, as identified by the Molecular Tumor Board | Baseline
Availability of targeted therapy from tumor material scored as category A, B, or C above or D) No target therapy available, or no genetic alterations found | Baseline
Overall survival | Number of days from enrollment to death, assessed up to 24 months
  Overall survival of patients in each cohort will be characterized using Kaplan-Meier plots and the two cohorts will be compared using a Cox model to control for age and sex.
Clinical response rate, assessed according to RECIST 1.1 criteria | Up to 24 months
  Response will be compared using logistic regression, adjusting for the same risk factors.
Incidence of adverse events | Up to 30 days after last dose of active treatment
  Categorized by grade and MedDRA preferred term.
Tumor-based genomics | Baseline
  Comparison of tumor-based genomics with peripheral-blood genomics will be carried out by comparing the list of genetic aberrations found in the two different samples (tumor vs ctDNA) and possible target drugs identified from each source. Agreement on success of profiling will be assessed using a kappa statistic.
Peripheral-blood genomics | Baseline
  Comparison of tumor-based genomics with peripheral-blood genomics will be carried out by comparing the list of genetic aberrations found in the two different samples (tumor vs ctDNA) and possible target drugs identified from each source. Agreement on success of profiling will be assessed using a kappa statistic.

CONTACTS AND LOCATIONS:
Overall Officials: James M Ford, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States